CLINICAL TRIAL: NCT06938308
Title: Comparison Between the I-gel and Protector Supraglottic Airway Devices in Patients Under General Anesthesia
Brief Title: Comparison Between the I-gel and Protector Supraglottic Airway Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nikolopoulou Maria Zozefin (Other)
Responsible Party: Sponsor-Investigator, Nikolopoulou Maria Zozefin, Anesthesiology Resident at Sismanoglio General Hospital, Sismanoglio General Hospital
Organization: Sismanoglio General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9254/10-04-2025
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-04

CONDITIONS: Airway Management; Learning Curve
Keywords: I-gel; Protector; learning curve; LMA; airway

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LMA Igel group (Active Comparator)
  Interventions: Device: LMA Igel
- LMA Protector group (Active Comparator)
  Interventions: Device: LMA Protector

INTERVENTIONS:
Device: LMA Igel — adults allocated to the LMA Igel group, an LMA Igel device will be inserted intraoperatively
  Arms: LMA Igel group
Device: LMA Protector — adults allocated to the LMA Protector group, an LMA Protector device will be inserted intraoperatively
  Arms: LMA Protector group

SUMMARY:
This study aims to compare the learning curves of two different laryngeal mask airway devices, by evaluating their placement in adult patients performed by anesthesiology residents

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Patients older than 18 years
* Procedures in supine and lithotomy position

Exclusion Criteria:

* Tumors or anatomical anomalies of the upper airway
* Known history of difficult intubation
* Limited mouth opening less than 2cm
* Decreased compliance of the lungs or the thoracic cage
* Need of mechanical ventilation after the surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
The time required for successful placement of the device | Measured from the moment the clinician picks up the LMA device after induction of general anesthesia until the appearance of the first capnography waveform on the monitor with a maximum duration of 60 seconds per attempt and up to three attempts allowed

SECONDARY OUTCOMES:
Documentation of adverse events during placement | During the placement attempt

CONTACTS AND LOCATIONS:
Locations (1):
- SismanoglioGH, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No